CLINICAL TRIAL: NCT06175000
Title: Maintenance Obinutuzumab for Primary Central Nervous System Lymphoma Complete or Partial Responders
Brief Title: Maintenance Obinutuzumab in Treating Patients With Central Nervous System Lymphoma Who Have Achieved a Complete or Partial Response
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHS-OB-PCNSL-01; ML29496 (Other: Genentech, Inc.); NCT02498951 (obsolete NCT alias)
Record Dates: First submitted 2023-06-28; First posted 2023-12-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — Mental Status and Dementia Tests; obinutuzumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (obinutuzumab (Experimental): Patients receive obinutuzumab IV on days 1 and 2 for the first cycle, and on day 1 for the subsequent cycles, and on day 1 for the subsequent cycles. Cycles repeat every 60 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Cognitive Assessment; Biological: Obinutuzumab; Other: Quality of Life Assessment
- Arm II (observation) (Active Comparator): Patients undergo observation for a total of 2 years.
  Interventions: Procedure: Cognitive Assessment; Other: Quality of Life Assessment

INTERVENTIONS:
Procedure: Cognitive Assessment — Ancillary studies to evaluate neurocognitive function at study entry and at 2 years after study entry.
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB (CD20); R7159; RO 5072759; RO-5072759; RO5072759
  Arms: Arm I (obinutuzumab
Other: Quality of Life Assessment — Ancillary studies to evaluate quality of life at study entry and at 2 years after study entry.

SUMMARY:
This randomized phase II trial studies how well obinutuzumab works as maintenance treatment in patients with central nervous system lymphoma who have achieved the disappearance of all signs of cancer in response to treatment (complete response) or a decrease in the size of a tumor, or in the extent of cancer in the body, in response to treatment (partial response). Immunotherapy with obinutuzumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of maintenance obinutuzumab on duration of response (partial response [PR] or complete response [CR]) in patients with CD20+ B-cell primary central nervous system lymphoma (PCNSL) who attain PR or CR to first-line treatment with high-dose methotrexate-based chemotherapy.

SECONDARY OBJECTIVES:

I. To evaluate overall survival after PR or CR (overall survival [OS]-PRCR). II. To evaluate neurocognitive function, quality of life, and neuroimaging as indicators of neurotoxicity.

III. Progression-free survival (PFS) and overall survival (OS) will be calculated.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (MAINTENANCE THERAPY): Patients receive obinutuzumab intravenously (IV) on days 1 and 2 for the first cycle, and on day 1 for the subsequent cycles. Cycles repeat every 60 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM II (OBSERVATION): Patients undergo observation for a total of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* CD20+ B-cell primary central nervous system lymphoma (PCNSL) confirmed at the time of diagnosis by histology, cytology, or immunocytochemistry from cerebrospinal fluid (CSF); diagnosis must be documented by pathology report.
* Must have undergone first-line treatment with a high-dose methotrexate-based chemotherapy regimen with or without brain radiotherapy; high-dose methotrexate is defined as >= 3 grams/m^2; methotrexate dose reduction for creatinine clearance < 100 ml/min is permitted
* Must be within 75 days of completion of first-line treatment regimen at the time of randomization; must have achieved objective response (PR or CR/unconfirmed complete response [CRu]) to first-line treatment
* Brain magnetic resonance imaging (MRI) documenting objective response must be obtained within 30 days before randomization
* If CSF was positive for lymphoma cells at diagnosis or during first-line treatment and/or a slit lamp examination was positive at diagnosis or during first-line treatment, then the CSF and vitreal studies must have been repeated and must have indicated CR; Note: CR requires complete disappearance of all enhancing abnormalities on gadolinium-enhanced MRI; if CSF was positive for lymphoma cells at diagnosis or during first-line treatment and/or slit lamp examination was positive at diagnosis or during first-line treatment, then the CSF and vitreal studies must have been repeated and must have indicated CR; for CRu, some patients will have a small but persistent enhancing abnormality on MRI related to biopsy or focal hemorrhage; it is often difficult to ascertain whether this represents a residual nidus of tumor or scar tissue; if the abnormality does not change or slowly involutes without therapy and corticosteroids, it is reasonable to categorize as a CRu; at the time CR/CRu is determined, the patient should not have used corticosteroids for at least two weeks
* Karnofsky performance status (KPS) >= 60; Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2
* Signed informed consent form (ICF)
* Ability and willingness to comply with the requirements of the study protocol
* Total bilirubin < 3 x the upper limit of normal (ULN), ≤ 7 days before date of randomization
* Creatinine clearance > 30 mL/min (calculated according to institutional standards or using Cockcroft-Gault formula), ≤ 7 days before date of randomization
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 5 x ULN, ≤7 days before date of randomization
* Platelet ≤ 75,000 cells/mm^3, ≤ 7 days before date of randomization
* Hemoglobin > 9 g/dL, ≤ 7 days before date of randomization
* Absolute neutrophil count > 1.5 x 10^3 cells/mm^3, ≤ 7 days before date of randomization
* Surgically sterile or agree to use effective contraception using an adequate measure of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly while receiving obinutuzumab and >= 18 months after the last dose of obinutuzumab for women, and 180 days after the last dose of obinutuzumab for men

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Clinical evidence of extra-central nervous system (CNS) (systemic) non-Hodgkin lymphoma
* Known hypersensitivity to any of the study drugs
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are generally eligible; patients with a malignancy that has been treated, but not with curative intent, will also be excluded, unless the malignancy has been in remission without treatment for >= 2 years prior to randomization
* Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks prior to study randomization
* Major surgery within 4 weeks prior to study randomization
* Known infection with human immunodeficiency virus (HIV)
* Positive hepatitis serologies:
* Hepatitis B (HBV): patients with positive serology for hepatitis B defined as positivity for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (anti-HBc); patients who are positive for anti-HBc may be considered for inclusion in the study on a case-by-case basis if they are hepatitis B viral deoxyribonucleic acid (DNA) negative and are willing to undergo ongoing HBV DNA testing by real-time polymerase chain reaction (PCR); patients with positive serology may be referred to a hepatologist or gastroenterologist for appropriate monitoring and management
* Hepatitis C (HCV): patients with positive hepatitis C serology unless HCV ribonucleic acid (RNA) is confirmed negative and may be considered for inclusion in the study on a case-by-case basis
* Women who are pregnant or lactating
* Vaccination with a live vaccine a minimum of 4 weeks prior to study randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Partial response (PR) or complete response (CR) duration | From the date of brain magnetic resonance imaging (MRI) after completion of first-line treatment which confirms PR or CR, to disease progression or death, assessed up to 2 years
  PR or CR duration will be assessed using Kaplan-Meier product limit estimates and compared between patients with maintenance versus without obinutuzumab maintenance using the log-rank test. In addition, the Cox proportional hazard model will be used to estimate hazard ratios.

SECONDARY OUTCOMES:
Overall survival (OS) after CR | From the date of brain MRI after completion of first-line treatment which confirms PR or CR, to death, assessed up to 2 years
  OS after PR or CR will be assessed using Kaplan-Meier product limit estimates and compared between patients with maintenance versus without obinutuzumab maintenance using the log-rank test. In addition, the Cox proportional hazard model will be used to estimate hazard ratios.
Neurocognitive function - Wechsler Adult Intelligence Scale | Up to 2 years
  Will be measured by the Wechsler Adult Intelligence Scale. Scale range 0 to 16 Forward; 0 to 14 Backward. Higher the score means better outcome. Longitudinal data of neurocognitive function will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Quality of life (QOL) - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Brain Neoplasm 20-item | Up to 2 years
  Will be measured by the European Organization for Research and Treatment of Cancer Quality of Life Brain Cancer Module-20 (EORTC QLQ-BN20) questionnaire. Scale 20 to 80 points. Higher score means worse outcome. Longitudinal data of QOL will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Progression free survival (PFS) | From the start date of first-line primary central nervous system lymphoma (PCNSL) treatment to disease progression or death, assessed up to 2 years
  PFS will be assessed using Kaplan-Meier product limit estimates and compared between patients with obinutuzumab maintenance versus without maintenance using the log-rank test. Longitudinal data of neurocognitive function and QOL will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Overall survival | From the start date of first-line PCNSL treatment to death, assessed up to 2 years.
  OS will be assessed using Kaplan-Meier product limit estimates and compared between patients with obinutuzumab maintenance versus without maintenance using the log-rank test. Longitudinal data of neurocognitive function and QOL will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Neurocognitive function - Hopkins Verbal Learning Test-Revised | Up to 2 years
  Will be measured by the Hopkins Verbal Learning Test-Revised. Test evaluates total recall, delayed recall, percent of retention, and recognition. Higher score means better outcome. Longitudinal data of neurocognitive function will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Neurocognitive function - Grooved Pegboard Test | Up to 2 years
  Will be measured by the Grooved Pegboard Test. Scale 0 seconds to time of completion in minutes and seconds. Higher time to completion means worse outcome. Longitudinal data of neurocognitive function will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Neurocognitive function - Trail Making Test | Up to 2 years
  Will be measured by the Trail Making Test. Scale Part A: 0 seconds to 100 seconds (time of greater than 100 seconds discontinues the test. Scale Part B: 0 seconds to 300 seconds (time of greater than 300 seconds discontinues the test. Number of errors recorded. Higher time to completion and greater number of errors means worse outcome. Longitudinal data of neurocognitive function will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Neurocognitive function - Brief Test of Attention | Up to 2 years
  Will be measured by the Trail Making Test. Scale 0 to 20 points. Higher score mean better outcome. Longitudinal data of neurocognitive function will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.
Quality of life (QOL) - European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30-item | Up to 2 years
  Will be measured by the European Organization for Research and Treatment of Cancer Quality of Life Core 30-item (EORTC QLQ-C30) questionnaire. Scale 30 to 126 points. Higher score means worse outcome. Longitudinal data of QOL will be analyzed using a linear mixed model and toxicity indicators will be assessed using a chi-square or exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Ambady, MD, Principal Investigator — Providence Health & Services
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Health & Services; Providence Neurological Specialties, Portland, Oregon
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Vermont, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Ivy Center for Advanced Brain Tumor Treatment; Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No